CLINICAL TRIAL: NCT03593772
Title: Mission Reconnect: Delivering a Mobile and Web Based Self Directed Complementary and Integrative Health Program to Veterans and Their Partners to Manage Pain and PTSD
Brief Title: Mission Reconnect-Veterans and Their Partners to Manage Pain and PTSD (MR)
Acronym: MR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D2775-R
Record Dates: First submitted 2018-05-22; First posted 2018-07-20 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: PTSD; Chronic Musculoskeletal Pain
Keywords: chronic pain; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This research study will evaluate a CIH intervention to manage pain and PTSD related outcomes within a bio-psychosocial framework. The proposed intervention, Mission Reconnect (MR), a user-driven, dyadic, self-care management program delivered online and by mobile app that has previously shown to be effective in a non-clinically defined community-based Veteran/military population.
Masking Description: There are no masked roles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment arm - Veteran (Active Comparator): Treatment Arm: MR is an user-driven, dyadic, self-care management program developed with National Institute of Mental Health (NIMH) funding (R43/44) for use by Veterans and their selected partners, individually or together, to reduce pain and distress and support physical, mental, and relationship health. MR was designed for Veterans who face obstacles accessing formal mental health services. It can also be used to complement formal services. MR is a patient-centered intervention, allowing users to determine the pace at which to proceed in each program component. MR Content. The program provides video and audio instruction in a set of 11 evidence-based wellness.
  Interventions: Behavioral: Mission Reconnect
- Control arm - Veteran (No Intervention): Usual Care Waitlist Control Arm: For ethical reasons, this study will use a waitlist control arm to ultimately provide all participants exposure to the MR intervention. Dyads in the control arm will participate in all assessments like those in the treatment group, however, they will be asked to agree to not access the public web site during their participation. Wait-list control participants will be instructed to seek advice about treatment from their providers. Other than this initial advice, there will be no attempt by study personnel to influence condition management unless an issue (i.e., suicidal ideation) arises. The control condition will account for potential temporal effects that occur from passage of time (brief), and expectation effects associated with anticipation of MR participation. The control group will receive access to MR after they complete data collection.
- Treatment arm - Partner (Experimental): Treatment Arm: MR is an user-driven, dyadic, self-care management program developed with NIMH funding (R43/44) for use by Veterans and their selected partners, individually or together, to reduce pain and distress and support physical, mental, and relationship health. MR was designed for Veterans who face obstacles accessing formal mental health services. It can also be used to complement formal services. MR is a patient-centered intervention, allowing users to determine the pace at which to proceed in each program component. MR Content. The program provides video and audio instruction in a set of 11 evidence-based wellness.
  Interventions: Behavioral: Mission Reconnect
- Control arm - Partner (No Intervention): Usual Care Waitlist Control Arm: For ethical reasons, this study will use a waitlist control arm to ultimately provide all participants exposure to the MR intervention. Dyads in the control arm will participate in all assessments like those in the treatment group, however, they will be asked to agree to not access the public web site during their participation. Wait-list control participants will be instructed to seek advice about treatment from their providers. Other than this initial advice, there will be no attempt by study personnel to influence condition management unless an issue (i.e., suicidal ideation) arises. The control condition will account for potential temporal effects that occur from passage of time (brief), and expectation effects associated with anticipation of MR participation. The control group will receive access to MR after they complete data collection.

INTERVENTIONS:
Behavioral: Mission Reconnect — This four-year randomized controlled trial with one intervention arm and one wait-list control arm will utilize mixed methods to evaluate the effectiveness and perceived value of the MR program in relation to physical and psychological symptoms, global health, and social outcomes.
  Arms: Treatment arm - Partner; Treatment arm - Veteran

SUMMARY:
This project is responsive to Rehabilitation Research and Development's (RR&D) current special areas of interest for non-pharmacological activity-based interventions for chronic pain impacting pain reduction, function and quality of life. This project aligns with the VA mandate for complementary and integrative health (CIH) care for Veterans and their families. CIH complements traditional care for Veterans managing chronic conditions, such as chronic pain and PTSD. Mission Reconnect (MR) is a user-driven, dyadic, CIH self-care management program delivered remotely that teaches techniques the Veteran/partner dyad can use to reduce pain, anxiety and stress, promote well-being and improve relationship quality. The research goal is to evaluate MR as an approach to manage chronic pain and PTSD symptoms, for potential subsequent implementation. This study will possibly provide a model for establishing remote access and sustainable implementation of CIH within VA.

DETAILED DESCRIPTION:
Chronic pain is one of the most prevalent medical conditions in the Veteran population. Pain often presents with comorbid conditions, specifically post-traumatic stress disorder (PTSD). Comorbid chronic pain and PTSD significantly impact the quality of life of Veterans and their families. Multi-faceted therapies leveraging complementary and integrative health (CIH) are mandated within VA to complement clinical practice guidelines improve Veterans' quality of life and ability to function. This research will evaluate a CIH intervention to manage pain and PTSD related outcomes within a bio-psychosocial framework. The proposed intervention, Mission Reconnect (MR), a user-driven, dyadic, self-care management program delivered online and by mobile app that has previously shown to be effective in a non-clinically defined community-based Veteran/military population. This research is needed to test MR's effects in a clinically defined population as a complement to clinical services to assess for potential subsequent implementation within the Department of Veterans Affairs (VA).

This proposal resubmission is responsive to Veterans' reported desire for CIH and several VA initiatives, including RR&D's current special areas of interest for non-pharmacological activity-based interventions for chronic pain impacting pain reduction, function and quality of life. The VA Secretary of Health Strategic Priorities and the emerging VA Whole Health Program identify access to CIH for pain and self-care management as a priority to achieve optimal Veteran health. To be responsive to these priorities the 2016 VA State-of-the-Art Conference (SOTA) and Comprehensive Addiction Recovery Act (CARA) mandated VA's commitment to conduct rigorous research to integrate non-pharmacological and CIH approaches into care, with emphasis on pain management. This proposal is also responsive to the VA's Opioid Safety Initiative (OSI) and Pain Care Mission which prioritize the need for nonpharmacological treatment options for pain. The short-term goal of this study is to determine the effects of MR on (1) chronic pain, PTSD and related outcomes and (2) relationship outcomes for Veterans and their partners. The long-term goal is to determine the effectiveness and sustainability of using CIH self-care management programs like MR to improve outcomes for Veterans with chronic pain and PTSD, and their partners. The investigators propose a four-year mixed-methods randomized controlled trial of MR with two arms (treatment & wait-list control) in a clinical sample of Veterans with comorbid pain and PTSD, and their partners (e.g., spouse). The specific aims are to: (Aim 1) Determine MR effectiveness for physical (pain, sleep), PTSD (intrusion, arousal, avoidance, numbing), and psychological (depression, stress, anxiety) symptoms, and global health (quality of life); (Aim 2) Determine MR effectiveness for social (relationship satisfaction, compassion for self/others) outcomes among Veterans and their partners; and (Aim 3) Describe Veteran and partner perceived value of MR in a sub-sample of participants. The sample will consist of Veteran and partner dyads (N = 336) at the Ann Arbor, Puget Sound, and Tampa VA facilities. Aim 1 & 2 data collection will include self-report assessment of 4-data points over a 4-month period to evaluate physical, psychological, and social outcomes. Eight weekly reports will also be collected for the first two months of MR use to assess MR utilization, and pain and stress levels. Aim 3 data collection will include telephone interviews from a randomly selected sub-sample of MR treatment group dyads (n = 42) to examine MR user experiences and their suggestions making MR useful for Veterans and their partners.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking Veterans with chronic musculoskeletal pain.
* Veteran is considered to have chronic musculoskeletal pain if he or she meeting either of two validated criteria:

  * (1) Having 2+ occurrences of any of targeted musculoskeletal ICD-9-CM codes "likely to represent chronic pain" recorded at visits separated by at least 30 days within past six months
  * (2) Having high impact chronic pain = 2+ occurrences of targeted musculoskeletal ICD-9-CM codes separated by at least 30 days within the past six months previous to study recruitment and two or more pain scores greater than or equal to 4 separated by at least 30 days within past six months.
* For pain scores, the investigators will use the 0-10 numeric pain rating scale that is routinely collected at the VA.

  * The investigators will count two ICD-9-CM codes or pain scores recorded on the same day as one code/score.
  * Veteran is considered to have PTSD if he or she has a flag in his/her record indicating confirmed condition by the VA Compensation and Benefits program, has at least two outpatient visits in the year with the primary diagnosis being listed as PTSD (ICD-9-CM code 309.81) and/or had PTSD listed on the problem list], Veteran must also have PTSD (defined by PTSD diagnosis-ICD-9-CM 309.81), the ability to access and use an electronic platform (e.g. Mobile device, internet, DVD) for MR delivery, with a willing partner to also participate in the study and MR program.

Exclusion Criteria:

* Moderate to severe traumatic brain injury (TBI)
* Diagnosis or documented treatment for psychosis in previous 6 months
* Currently in substance use disorder treatment
* Non-English speaking
* Visual, hearing, cognitive impairment that prevent participation or ability to consent
* And/or lack of access to internet service
* These individuals will be excluded due to medical, language, and technology access issues that would prevent safe and full study participation.
* Pain and PTSD treatment will not be factored as an inclusion/exclusion criteria but will be evaluated as covariates.
* Potential participants who screen for aggression or violence will also be excluded from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolie N. Haun, PhD MS BS, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (3):
- United States (3):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Dissemination efforts will be led by Drs. Haun, French, and Fowler, in cooperation with VA operational [e.g. Office of Patient Centered Care and Cultural Transformation (OPCCCT) and Office of Connected Care (OCC)], and clinical stakeholders (e.g. mental health and pain clinicians). The investigators will publish findings in peer-reviewed journals and present findings at national and international meetings including Medicine 2.0, the international conference for internet-based health research (Haun) and Association of Military Surgeons of the United States (AMSUS) Annual Continuing Education Meeting. Dissemination activities will inform Veterans Health Administration (VHA) operational initiatives and clinical practice. The deployment of Whole Health models of care nationally will provide a natural setting for dissemination. The Tampa VEC will support dissemination efforts to Veterans, their families, and to Veteran Service Organizations.

REFERENCES:
- [Background] Kip KE, Rosenzweig L, Hernandez DF, Shuman A, Diamond DM, Girling SA, Sullivan KL, Wittenberg T, Witt AM, Lengacher CA, Anderson B, McMillan SC. Accelerated Resolution Therapy for treatment of pain secondary to symptoms of combat-related posttraumatic stress disorder. Eur J Psychotraumatol. 2014 May 7;5. doi: 10.3402/ejpt.v5.24066. eCollection 2014. PMID 24959325
- [Background] Goulet JL, Kerns RD, Bair M, Becker WC, Brennan P, Burgess DJ, Carroll CM, Dobscha S, Driscoll MA, Fenton BT, Fraenkel L, Haskell SG, Heapy AA, Higgins DM, Hoff RA, Hwang U, Justice AC, Piette JD, Sinnott P, Wandner L, Womack JA, Brandt CA. The musculoskeletal diagnosis cohort: examining pain and pain care among veterans. Pain. 2016 Aug;157(8):1696-1703. doi: 10.1097/j.pain.0000000000000567. PMID 27023420
- [Background] Seal KH, Shi Y, Cohen G, Cohen BE, Maguen S, Krebs EE, Neylan TC. Association of mental health disorders with prescription opioids and high-risk opioid use in US veterans of Iraq and Afghanistan. JAMA. 2012 Mar 7;307(9):940-7. doi: 10.1001/jama.2012.234. PMID 22396516
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Sharp TJ, Harvey AG. Chronic pain and posttraumatic stress disorder: mutual maintenance? Clin Psychol Rev. 2001 Aug;21(6):857-77. doi: 10.1016/s0272-7358(00)00071-4. PMID 11497210
- [Background] Tsang A, Von Korff M, Lee S, Alonso J, Karam E, Angermeyer MC, Borges GL, Bromet EJ, Demytteneare K, de Girolamo G, de Graaf R, Gureje O, Lepine JP, Haro JM, Levinson D, Oakley Browne MA, Posada-Villa J, Seedat S, Watanabe M. Common chronic pain conditions in developed and developing countries: gender and age differences and comorbidity with depression-anxiety disorders. J Pain. 2008 Oct;9(10):883-91. doi: 10.1016/j.jpain.2008.05.005. Epub 2008 Jul 7. PMID 18602869
- [Background] Clark ME, Walker RL, Gironda RJ, Scholten JD. Comparison of pain and emotional symptoms in soldiers with polytrauma: unique aspects of blast exposure. Pain Med. 2009 Apr;10(3):447-55. doi: 10.1111/j.1526-4637.2009.00590.x. PMID 19416436
- [Background] Smeeding SJ, Bradshaw DH, Kumpfer KL, Trevithick S, Stoddard GJ. Outcome evaluation of the Veterans Affairs Salt Lake City Integrative Health Clinic for Chronic Nonmalignant Pain. Clin J Pain. 2011 Feb;27(2):146-55. doi: 10.1097/AJP.0b013e3181f158e8. PMID 20842019
- [Background] Shi L, Liu J, Zhao Y. Comparative effectiveness in pain-related outcomes and health care utilizations between veterans with major depressive disorder treated with duloxetine and other antidepressants: a retrospective propensity score-matched comparison. Pain Pract. 2012 Jun;12(5):374-81. doi: 10.1111/j.1533-2500.2011.00495.x. Epub 2011 Sep 27. PMID 21951787
- [Background] Lang KP, Veazey-Morris K, Andrasik F. Exploring the role of insomnia in the relation between PTSD and pain in veterans with polytrauma injuries. J Head Trauma Rehabil. 2014 Jan-Feb;29(1):44-53. doi: 10.1097/HTR.0b013e31829c85d0. PMID 23835878
- [Background] Kupersmith J, Lew HL, Ommaya AK, Jaffee M, Koroshetz WJ. Traumatic brain injury research opportunities: results of Department of Veterans Affairs Consensus Conference. J Rehabil Res Dev. 2009;46(6):vii-xvi. doi: 10.1682/jrrd.2009.06.0079. No abstract available. PMID 20104393
- [Background] Bosco MA, Murphy JL, Clark ME. Chronic pain and traumatic brain injury in OEF/OIF service members and Veterans. Headache. 2013 Oct;53(9):1518-22. doi: 10.1111/head.12172. Epub 2013 Jul 12. PMID 23848062
- [Background] Schnurr PP, Lunney CA. Work-related outcomes among female veterans and service members after treatment of posttraumatic stress disorder. Psychiatr Serv. 2012 Nov;63(11):1072-9. doi: 10.1176/appi.ps.201100415. PMID 22983600
- [Background] Westanmo A, Marshall P, Jones E, Burns K, Krebs EE. Opioid Dose Reduction in a VA Health Care System--Implementation of a Primary Care Population-Level Initiative. Pain Med. 2015 May;16(5):1019-26. doi: 10.1111/pme.12699. Epub 2015 Feb 3. PMID 25645538
- [Background] Capehart B, Bass D. Review: managing posttraumatic stress disorder in combat veterans with comorbid traumatic brain injury. J Rehabil Res Dev. 2012;49(5):789-812. doi: 10.1682/jrrd.2011.10.0185. PMID 23015586
- [Background] Engel GL. The clinical application of the biopsychosocial model. Am J Psychiatry. 1980 May;137(5):535-44. doi: 10.1176/ajp.137.5.535. PMID 7369396
- [Background] Gatchel RJ, Peng YB, Peters ML, Fuchs PN, Turk DC. The biopsychosocial approach to chronic pain: scientific advances and future directions. Psychol Bull. 2007 Jul;133(4):581-624. doi: 10.1037/0033-2909.133.4.581. PMID 17592957
- [Background] Geisser ME, Roth RS, Bachman JE, Eckert TA. The relationship between symptoms of post-traumatic stress disorder and pain, affective disturbance and disability among patients with accident and non-accident related pain. Pain. 1996 Aug;66(2-3):207-14. doi: 10.1016/0304-3959(96)03038-2. PMID 8880842
- [Background] Raichle KA, Romano JM, Jensen MP. Partner responses to patient pain and well behaviors and their relationship to patient pain behavior, functioning, and depression. Pain. 2011 Jan;152(1):82-88. doi: 10.1016/j.pain.2010.09.015. Epub 2010 Oct 13. PMID 20947249
- [Background] Verbosky SJ, Ryan DA. Female partners of Vietnam veterans: stress by proximity. Issues Ment Health Nurs. 1988;9(1):95-104. doi: 10.3109/01612848809140912. No abstract available. PMID 3356550
- [Background] Keefe FJ, Caldwell DS, Baucom D, Salley A, Robinson E, Timmons K, Beaupre P, Weisberg J, Helms M. Spouse-assisted coping skills training in the management of osteoarthritic knee pain. Arthritis Care Res. 1996 Aug;9(4):279-91. doi: 10.1002/1529-0131(199608)9:43.0.co;2-6. PMID 8997917
- [Background] Abbasi M, Dehghani M, Keefe FJ, Jafari H, Behtash H, Shams J. Spouse-assisted training in pain coping skills and the outcome of multidisciplinary pain management for chronic low back pain treatment: a 1-year randomized controlled trial. Eur J Pain. 2012 Aug;16(7):1033-43. doi: 10.1002/j.1532-2149.2011.00097.x. Epub 2012 Jan 19. PMID 22337646
- [Background] Baucom DH, Shoham V, Mueser KT, Daiuto AD, Stickle TR. Empirically supported couple and family interventions for marital distress and adult mental health problems. J Consult Clin Psychol. 1998 Feb;66(1):53-88. doi: 10.1037//0022-006x.66.1.53. PMID 9489262
- [Background] Monson CM, Macdonald A, Brown-Bowers A. Couple/family therapy for posttraumatic stress disorder: review to facilitate interpretation of VA/DOD Clinical Practice Guideline. J Rehabil Res Dev. 2012;49(5):717-28. doi: 10.1682/jrrd.2011.09.0166. PMID 23015582
- [Background] Church D, Brooks AJ. CAM and energy psychology techniques remediate PTSD symptoms in veterans and spouses. Explore (NY). 2014 Jan-Feb;10(1):24-33. doi: 10.1016/j.explore.2013.10.006. Epub 2013 Oct 17. PMID 24439093
- [Background] Kahn JR, Collinge W, Soltysik R. Post-9/11 Veterans and Their Partners Improve Mental Health Outcomes with a Self-directed Mobile and Web-based Wellness Training Program: A Randomized Controlled Trial. J Med Internet Res. 2016 Sep 27;18(9):e255. doi: 10.2196/jmir.5800. PMID 27678169
- [Background] Denneson LM, Corson K, Dobscha SK. Complementary and alternative medicine use among veterans with chronic noncancer pain. J Rehabil Res Dev. 2011;48(9):1119-28. doi: 10.1682/jrrd.2010.12.0243. PMID 22234716
- [Background] Herman PM, Sorbero ME, Sims-Columbia AC. Complementary and Alternative Medicine Services in the Military Health System. J Altern Complement Med. 2017 Nov;23(11):837-843. doi: 10.1089/acm.2017.0236. Epub 2017 Oct 17. PMID 29039681
- [Background] Peterson K, Anderson J, Ferguson L, Mackey K. Evidence Brief: The Comparative Effectiveness of Selected Complementary and Integrative Health (CIH) Interventions for Preventing or Reducing Opioid Use in Adults with Chronic Neck, Low Back, and Large Joint Pain [Internet]. Washington (DC): Department of Veterans Affairs (US); 2016 Apr. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK409241/ PMID 28102991
- [Background] Haun JN, Graham-Pole J, Shortley B. Children with cancer and blood diseases experience positive physical and psychological effects from massage therapy. Int J Ther Massage Bodywork. 2009 Jun 29;2(2):7-14. doi: 10.3822/ijtmb.v2i2.12. PMID 21589728
- [Background] Cherkin DC, Eisenberg D, Sherman KJ, Barlow W, Kaptchuk TJ, Street J, Deyo RA. Randomized trial comparing traditional Chinese medical acupuncture, therapeutic massage, and self-care education for chronic low back pain. Arch Intern Med. 2001 Apr 23;161(8):1081-8. doi: 10.1001/archinte.161.8.1081. PMID 11322842
- [Background] Moyer CA, Rounds J, Hannum JW. A meta-analysis of massage therapy research. Psychol Bull. 2004 Jan;130(1):3-18. doi: 10.1037/0033-2909.130.1.3. PMID 14717648
- [Background] Tsao JC. Effectiveness of massage therapy for chronic, non-malignant pain: a review. Evid Based Complement Alternat Med. 2007 Jun;4(2):165-79. doi: 10.1093/ecam/nel109. Epub 2007 Feb 5. PMID 17549233
- [Background] Crawford C, Boyd C, Paat CF, Price A, Xenakis L, Yang E, Zhang W; Evidence for Massage Therapy (EMT) Working Group. The Impact of Massage Therapy on Function in Pain Populations-A Systematic Review and Meta-Analysis of Randomized Controlled Trials: Part I, Patients Experiencing Pain in the General Population. Pain Med. 2016 Jul 1;17(7):1353-1375. doi: 10.1093/pm/pnw099. PMID 27165971
- [Background] Sharpe PA, Williams HG, Granner ML, Hussey JR. A randomised study of the effects of massage therapy compared to guided relaxation on well-being and stress perception among older adults. Complement Ther Med. 2007 Sep;15(3):157-63. doi: 10.1016/j.ctim.2007.01.004. Epub 2007 Feb 20. PMID 17709060
- [Background] Moraska A, Pollini RA, Boulanger K, Brooks MZ, Teitlebaum L. Physiological adjustments to stress measures following massage therapy: a review of the literature. Evid Based Complement Alternat Med. 2010 Dec;7(4):409-18. doi: 10.1093/ecam/nen029. Epub 2008 May 7. PMID 18955340
- [Background] Haun J, Patel N, Schwartz G, Ritenbaugh C. Evaluating the use of gas discharge visualization to measure massage therapy outcomes. J Complement Integr Med. 2015 Sep;12(3):231-9. doi: 10.1515/jcim-2014-0014. PMID 26087069
- [Background] Stephenson KR, Simpson TL, Martinez ME, Kearney DJ. Changes in Mindfulness and Posttraumatic Stress Disorder Symptoms Among Veterans Enrolled in Mindfulness-Based Stress Reduction. J Clin Psychol. 2017 Mar;73(3):201-217. doi: 10.1002/jclp.22323. Epub 2016 May 6. PMID 27152480
- [Background] Garland EL, Manusov EG, Froeliger B, Kelly A, Williams JM, Howard MO. Mindfulness-oriented recovery enhancement for chronic pain and prescription opioid misuse: results from an early-stage randomized controlled trial. J Consult Clin Psychol. 2014 Jun;82(3):448-459. doi: 10.1037/a0035798. Epub 2014 Feb 3. PMID 24491075
- [Background] Serpa JG, Taylor SL, Tillisch K. Mindfulness-based stress reduction (MBSR) reduces anxiety, depression, and suicidal ideation in veterans. Med Care. 2014 Dec;52(12 Suppl 5):S19-24. doi: 10.1097/MLR.0000000000000202. PMID 25397818
- [Background] Nash WP, Watson PJ. Review of VA/DOD Clinical Practice Guideline on management of acute stress and interventions to prevent posttraumatic stress disorder. J Rehabil Res Dev. 2012;49(5):637-48. doi: 10.1682/jrrd.2011.10.0194. PMID 23015576
- [Background] Elwy AR, Johnston JM, Bormann JE, Hull A, Taylor SL. A systematic scoping review of complementary and alternative medicine mind and body practices to improve the health of veterans and military personnel. Med Care. 2014 Dec;52(12 Suppl 5):S70-82. doi: 10.1097/MLR.0000000000000228. PMID 25397827
- [Background] Engel GL. The need for a new medical model: a challenge for biomedicine. Science. 1977 Apr 8;196(4286):129-36. doi: 10.1126/science.847460.
- [Background] Cohen S, Wills TA. Stress, social support, and the buffering hypothesis. Psychol Bull. 1985 Sep;98(2):310-57. No abstract available. PMID 3901065
- [Background] Collinge W, Kahn J, Soltysik R. Promoting reintegration of National Guard veterans and their partners using a self-directed program of integrative therapies: a pilot study. Mil Med. 2012 Dec;177(12):1477-85. doi: 10.7205/milmed-d-12-00121. PMID 23397692
- [Background] Tian TY, Zlateva I, Anderson DR. Using electronic health records data to identify patients with chronic pain in a primary care setting. J Am Med Inform Assoc. 2013 Dec;20(e2):e275-80. doi: 10.1136/amiajnl-2013-001856. Epub 2013 Jul 31. PMID 23904323
- [Background] Sandelowski M. Sample size in qualitative research. Res Nurs Health. 1995 Apr;18(2):179-83. doi: 10.1002/nur.4770180211. PMID 7899572
- [Background] Ritenbaugh C, Nichter M, Nichter MA, Kelly KL, Sims CM, Bell IR, Castaneda HM, Elder CR, Koithan MS, Sutherland EG, Verhoef MJ, Warber SL, Coons SJ. Developing a patient-centered outcome measure for complementary and alternative medicine therapies I: defining content and format. BMC Complement Altern Med. 2011 Dec 29;11:135. doi: 10.1186/1472-6882-11-135. PMID 22206345
- [Background] Thompson JJ, Kelly KL, Ritenbaugh C, Hopkins AL, Sims CM, Coons SJ. Developing a patient-centered outcome measure for complementary and alternative medicine therapies II: refining content validity through cognitive interviews. BMC Complement Altern Med. 2011 Dec 29;11:136. doi: 10.1186/1472-6882-11-136. PMID 22206409
- [Background] Corrigan JD, Bogner J. Initial reliability and validity of the Ohio State University TBI Identification Method. J Head Trauma Rehabil. 2007 Nov-Dec;22(6):318-29. doi: 10.1097/01.HTR.0000300227.67748.77. PMID 18025964
- [Background] Busija L, Pausenberger E, Haines TP, Haymes S, Buchbinder R, Osborne RH. Adult measures of general health and health-related quality of life: Medical Outcomes Study Short Form 36-Item (SF-36) and Short Form 12-Item (SF-12) Health Surveys, Nottingham Health Profile (NHP), Sickness Impact Profile (SIP), Medical Outcomes Study Short Form 6D (SF-6D), Health Utilities Index Mark 3 (HUI3), Quality of Well-Being Scale (QWB), and Assessment of Quality of Life (AQoL). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S383-412. doi: 10.1002/acr.20541. No abstract available. PMID 22588759
- [Background] Polomano RC, Galloway KT, Kent ML, Brandon-Edwards H, Kwon KN, Morales C, Buckenmaier C' 3rd. Psychometric Testing of the Defense and Veterans Pain Rating Scale (DVPRS): A New Pain Scale for Military Population. Pain Med. 2016 Aug;17(8):1505-19. doi: 10.1093/pm/pnw105. Epub 2016 Jun 6. PMID 27272528
- [Background] Clark ME, Gironda RJ, Young RW. Development and validation of the Pain Outcomes Questionnaire-VA. J Rehabil Res Dev. 2003 Sep-Oct;40(5):381-95. doi: 10.1682/jrrd.2003.09.0381. PMID 15080223
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Ten Have TR, Normand SL, Marcus SM, Brown CH, Lavori P, Duan N. Intent-to-Treat vs. Non-Intent-to-Treat Analyses under Treatment Non-Adherence in Mental Health Randomized Trials. Psychiatr Ann. 2008 Dec;38(12):772-783. doi: 10.3928/00485713-20081201-10. No abstract available. PMID 20717484
- [Result] Lew HL, Otis JD, Tun C, Kerns RD, Clark ME, Cifu DX. Prevalence of chronic pain, posttraumatic stress disorder, and persistent postconcussive symptoms in OIF/OEF veterans: polytrauma clinical triad. J Rehabil Res Dev. 2009;46(6):697-702. doi: 10.1682/jrrd.2009.01.0006. PMID 20104399
- [Derived] Haun JN, Fowler CA, Venkatachalam HH, Alman AC, Ballistrea LM, Schneider T, Benzinger RC, Melillo C, Alexander NB, Klanchar SA, Lapcevic WA, Bair MJ, Taylor SL, Murphy JL, French DD. Outcomes of a Remotely Delivered Complementary and Integrative Health Partnered Intervention to Improve Chronic Pain and Posttraumatic Stress Disorder Symptoms: Randomized Controlled Trial. J Med Internet Res. 2024 Oct 18;26:e57322. doi: 10.2196/57322. PMID 39422992
- [Derived] Haun JN, Venkatachalam HH, Fowler CA, Alman AC, Ballistrea LM, Schneider T, Benzinger RC, Melillo C, Alexander NB, Klanchar SA, Lapcevic W, French DD. Mobile and Web-Based Partnered Intervention to Improve Remote Access to Pain and Posttraumatic Stress Disorder Symptom Management: Recruitment and Attrition in a Randomized Controlled Trial. J Med Internet Res. 2023 Oct 3;25:e49678. doi: 10.2196/49678. PMID 37788078
- [Derived] Haun JN, Ballistrea LM, Melillo C, Standifer M, Kip K, Paykel J, Murphy JL, Fletcher CE, Mitchinson A, Kozak L, Taylor SL, Glynn SM, Bair M. A Mobile and Web-Based Self-Directed Complementary and Integrative Health Program for Veterans and Their Partners (Mission Reconnect): Protocol for a Mixed-Methods Randomized Controlled Trial. JMIR Res Protoc. 2019 May 13;8(5):e13666. doi: 10.2196/13666. PMID 31094345
- See also: ATLAS.ti: The Qualitative Data Analysis Software — http://www.atlasti.com/.
- See also: Statistical Analysis Software, SAS/STAT | SAS — http://www.sas.com/technologies/analytics/statistics/stat/index.html.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Instruments may be administered to different individuals at different timepoints. We consented 196 Veterans (Vs) to the Treatment arm (Tx) & 168 Vs to the Waitlist-control arm (WC). Some Partners (Ps) withdrew & new Ps were added to the study. We consented 198 Ps to Tx, & 168 Ps to WC. We have Baseline data for 141 Vs (Tx), 136 Vs (WC), 137 Ps (Tx), & 133 Ps (WC). Satisfaction/utilization were only obtained after Tx initiation. The n's are the number of individuals activated (133 Vs, 133 Ps).
Groups:
- Control Arm - Veteran; Control Arm - Partner: Usual Care Waitlist Control Arm: For ethical reasons, this study will use a waitlist control arm to ultimately provide all participants exposure to the MR intervention. Dyads in the control arm will participate in all assessments like those in the treatment group, however, they will be asked to agree to not access the public web site during their participation. Wait-list control participants will be instructed to seek advice about treatment from their providers. Other than this initial advice, there will be no attempt by study personnel to influence condition management unless an issue (i.e., suicidal ideation) arises. The control condition will account for potential temporal effects that occur from passage of time (brief), and expectation effects associated with anticipation of MR participation. The control group will receive access to MR after they complete data collection.
  Mission Reconnect: This four-year randomized controlled trial with one intervention arm and one wait-list control arm will utilize mixed methods to evaluate the effectiveness and perceived value of the MR program in relation to physical and psychological symptoms, global health, and social outcomes.
Period: Overall Study
Arm/Group | Treatment Arm - Veteran | Treatment Arm - Partner | Control Arm - Veteran | Control Arm - Partner
Started | 196 | 198 | 168 | 168
Completed Baseline Data Collection | 141 | 137 | 136 | 133
Activated in Protocol (Participants are activated if both Veteran and Partner register for the Mission Reconnect website, the partner acknowledges receipt of VA privacy practices, and both Veteran and Partner complete Baseline data collection activities.) | 133 | 133 | 133 | 133
Completed | 106 | 106 | 129 | 129
Not Completed | 90 | 92 | 39 | 39

BASELINE CHARACTERISTICS:
Population: Baseline data was collected from anyone who completed Baseline data collection.
Groups:
- Treatment Arm - Veteran; Treatment Arm - Partner: Treatment Arm: MR is an user-driven, dyadic, self-care management program developed with NIMH funding (R43/44) for use by Veterans and their selected partners, individually or together, to reduce pain and distress and support physical, mental, and relationship health. MR was designed for Veterans who face obstacles accessing formal mental health services. It can also be used to complement formal services. MR is a patient-centered intervention, allowing users to determine the pace at which to proceed in each program component. MR Content. The program provides video and audio instruction in a set of 11 evidence-based wellness.
  Mission Reconnect: This four-year randomized controlled trial with one intervention arm and one wait-list control arm will utilize mixed methods to evaluate the effectiveness and perceived value of the MR program in relation to physical and psychological symptoms, global health, and social outcomes.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm - Veteran | Treatment Arm - Partner | Control Arm - Veteran | Control Arm - Partner | Total
Number analyzed (Participants) | 196 | 198 | 168 | 168 | 730
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age was calculated at the time of when the participant was activated in the protocol (defined as when both the Veteran and the Partner completed all on-boarding activities). Participants where only one member completed data collection and on-boarding activities did not have an age calculated for them (n = 141 for the Treatment Arm, n = 136 for the Waitlist Control Arm). Population: The total number of individuals in each arm is the number of consents. We only rec'd Baseline data from 141 Veterans in the Mission Reconnect Arm, 137 Partners in the Mission Reconnect Arm, 136 Veterans in the Waitlist Control Arm, 133 Partners in the Waitlist Control Arm.
  Years
    number analyzed (Participants) | 141 | 137 | 136 | 133 | 547
    (all) | 55.80 (14.13) | 52.20 (13.72) | 57.28 (13.35) | 52.92 (14.57) | 56.54 (13.74)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 40 | 107 | 33 | 115 | 295
  Male | 100 | 29 | 103 | 17 | 249
  Other | 1 | 1 | 0 | 1 | 3
  No Data - Did not complete Baseline Data collection | 55 | 61 | 32 | 35 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 10 | 9 | 43
  Not Hispanic or Latino | 123 | 123 | 116 | 121 | 483
  Unknown or Not Reported | 60 | 64 | 42 | 38 | 204
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 3 | 1 | 1 | 0 | 5
  Asian (Chinese, Filipino, Japanese, Korean etc.) | 1 | 5 | 1 | 4 | 11
  Black and/or African American | 20 | 20 | 22 | 21 | 83
  Multiracial | 9 | 3 | 8 | 2 | 22
  White, Caucasian | 103 | 104 | 97 | 102 | 406
  Missing/Decline to Respond | 56 | 63 | 33 | 38 | 190
  Other | 4 | 2 | 6 | 1 | 13
Pain Outcomes Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Pain Range: 0 - 10 Mobility Range: 0 - 40 Activities of Daily Living Range: 0 - 40 Vitality Range: 0 - 30 Negative Affect Range: 0 - 50 Fear Range: 0 - 20 Total Range: 0-190. Higher Scores associated with more adverse pain-related patient reported outcomes. Population: Pain Outcomes Questionnaire was administered only to the Veterans. Only Demographics and Relationship measures were administered to the Partners. The total number of individuals in each arm is the number of consents. We only rec'd Baseline data from 141 Veterans in the Mission Reconnect Arm, 137 Partners in the Mission Reconnect Arm, 136 Veterans in the Waitlist Control Arm, 133 Partners in the Waitlist Control Arm.
  units on a scale
    Total POQ: number analyzed (Participants) | 141 | 0 | 136 | 0 | 277
    Total POQ | 103.50 (37.13) |  | 93.64 (33.08) |  | 98.66 (35.48)
    Pain: number analyzed (Participants) | 141 | 0 | 136 | 0 | 277
    Pain | 6.25 (1.91) |  | 6.07 (1.92) |  | 6.16 (1.91)
    Mobility: number analyzed (Participants) | 141 | 0 | 136 | 0 | 277
    Mobility | 21.63 (11.54) |  | 19.78 (10.78) |  | 20.72 (11.19)
    Activities of Daily Living: number analyzed (Participants) | 141 | 0 | 136 | 0 | 277
    Activities of Daily Living | 11.71 (11.24) |  | 10.07 (10.09) |  | 10.91 (10.70)
    Vitality: number analyzed (Participants) | 141 | 0 | 136 | 0 | 277
    Vitality | 20.60 (5.74) |  | 18.21 (5.71) |  | 19.43 (5.84)
    Negative Affect: number analyzed (Participants) | 141 | 0 | 136 | 0 | 277
    Negative Affect | 31.93 (11.59) |  | 28.61 (11.50) |  | 30.30 (11.64)
    Fear: number analyzed (Participants) | 141 | 0 | 136 | 0 | 277
    Fear | 11.38 (4.95) |  | 10.89 (4.88) |  | 11.14 (4.91)

OUTCOME MEASURES:

1. Primary Outcome: Pain Outcomes Questionnaire (POQ)
Description: 20-item questionnaire, used to assess pain, and pain-related subdomains, such as pain intensity, interference with activities, mobility, negative affect, vitality, and pain-related fear.
  Higher Scores associated with more adverse pain-related patient reported outcomes.
  Pain Range: 0 - 10 Mobility Range: 0 - 40 Activities of Daily Living Range: 0 - 40 Vitality Range: 0 - 30 Negative Affect Range: 0 - 50 Fear Range: 0 - 20 Total Range: 0-190
Time Frame: Baseline, month 1,2,4
Population: Multilinear model analyses were performed. Results provided are the Least Squares Mean and 95% C.I. for the two treatment arms. This is the least squares mean for the treatment variable averaged across all timepoints, after having controlled for other covariates. Instrument was administered only to Veterans activated in the protocol. Participants that opted out of responding were not included in the analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Treatment Arm: Treatment Arm: MR is an user-driven, dyadic, self-care management program developed with NIMH funding (R43/44) for use by Veterans and their selected partners, individually or together, to reduce pain and distress and support physical, mental, and relationship health. MR was designed for Veterans who face obstacles accessing formal mental health services. It can also be used to complement formal services. MR is a patient-centered intervention, allowing users to determine the pace at which to proceed in each program component. MR Content. The program provides video and audio instruction in a set of 11 evidence-based wellness.
  Mission Reconnect: This four-year randomized controlled trial with one intervention arm and one wait-list control arm will utilize mixed methods to evaluate the effectiveness and perceived value of the MR program in relation to physical and psychological symptoms, global health, and social outcomes.
- Control Arm: Usual Care Waitlist Control Arm: For ethical reasons, this study will use a waitlist control arm to ultimately provide all participants exposure to the MR intervention. Dyads in the control arm will participate in all assessments like those in the treatment group, however, they will be asked to agree to not access the public web site during their participation. Wait-list control participants will be instructed to seek advice about treatment from their providers. Other than this initial advice, there will be no attempt by study personnel to influence condition management unless an issue (i.e., suicidal ideation) arises. The control condition will account for potential temporal effects that occur from passage of time (brief), and expectation effects associated with anticipation of MR participation. The control group will receive access to MR after they complete data collection.
  Mission Reconnect: This four-year randomized controlled trial with one intervention arm and one wait-list control arm will utilize mixed methods to evaluate the effectiveness and perceived value of the MR program in relation to physical and psychological symptoms, global health, and social outcomes.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 141 | 136
Units on a scale
  Total POQ | 102.32 [96.6204 to 108.03] | 94.9863 [89.3230 to 100.65]
  Pain Rating | 6.2006 [5.8999 to 6.5014] | 6.1251 [5.8330 to 6.4173]
  Mobility | 21.4893 [19.7487 to 23.2298] | 20.2530 [18.5225 to 21.9835]
  Activities of Daily Living | 12.1675 [10.4442 to 13.8908] | 10.4716 [8.7829 to 12.1603]
  Vitality | 20.2433 [19.3959 to 21.0906] | 18.6968 [17.8919 to 19.5018]
  Negative Affect | 30.7769 [28.9694 to 32.5843] | 28.2654 [26.4939 to 30.0369]
  Fear | 11.5500 [10.8467 to 12.2533] | 11.1400 [10.4626 to 11.8174]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Analysis performed on Total POQ Score as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.05. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0535, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.04819, Standard Error of Mean 0.02482
Statistical Analysis 2: Comparison: Treatment Arm vs Control Arm; Analysis performed on Pain Rating as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.05. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.3729, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00163, Standard Error of Mean 0.001826
Statistical Analysis 3: Comparison: Treatment Arm vs Control Arm; Analysis performed on Mobility as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.05. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.4124, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00593, Standard Error of Mean 0.007228
Statistical Analysis 4: Comparison: Treatment Arm vs Control Arm; Analysis performed on Activities of Daily Living as outcome variable. Linear mixed models were constructed with fixed effects terms for treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test if the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.05. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.6442, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00432, Standard Error of Mean 0.009334
Statistical Analysis 5: Comparison: Treatment Arm vs Control Arm; Analysis performed on Vitality as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.05. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1641, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00898, Standard Error of Mean 0.006436
Statistical Analysis 6: Comparison: Treatment Arm vs Control Arm; Analysis performed on Neg. Affect as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.05. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0487, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.01952, Standard Error of Mean 0.009846
Statistical Analysis 7: Comparison: Treatment Arm vs Control Arm; Analysis performed on Fear as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.05. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1554, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00660, Standard Error of Mean 0.004644

2. Secondary Outcome: Pain, Stress and Tension Likert
Description: Three items will assess pain, stress and tension using a 0 to 5-point Likert-type scale.
  Higher Scores associated with more adverse patient reported outcomes. Pain Range: 0 - 5 Stress Range: 0 - 5 Tension Range: 0 - 5
Time Frame: Baseline, Week 1 - 8, Week 16
Population: Multilinear model analyses were performed. Results provided are the Least Squares Mean and 95% C.I. for the two treatment arms. This is the least squares mean for the treatment variable averaged across all timepoints, after having controlled for other covariates. Instrument was administered only to Veterans who had been activated in the protocol. Participants who opted out of responding to certain questions were not included in the analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 141 | 136
units on a scale
  Pain (on 5-point Likert Scale): number analyzed (Participants) | 140 | 136
  Pain (on 5-point Likert Scale) | 3.3904 [3.2548 to 3.5260] | 3.3230 [3.1909 to 3.4551]
  Stress (on 5-point Likert Scale): number analyzed (Participants) | 140 | 136
  Stress (on 5-point Likert Scale) | 3.1728 [3.0109 to 3.3348] | 3.0601 [2.9035 to 3.2168]
  Tension (on 5-point Likert Scale): number analyzed (Participants) | 140 | 136
  Tension (on 5-point Likert Scale) | 3.4061 [3.2634 to 3.5487] | 3.2474 [3.1093 to 3.3855]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Analysis performed on Pain as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1924, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00113, Standard Error of Mean 0.000863
Statistical Analysis 2: Comparison: Treatment Arm vs Control Arm; Analysis performed on Stress as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1002, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00190, Standard Error of Mean 0.001152
Statistical Analysis 3: Comparison: Treatment Arm vs Control Arm; Analysis performed on Tension as the outcome variable. Linear mixed models were constructed with fixed effects terms for the treatment group (MR vs. WC), time (continuous), and a treatment group x time interaction term to test whether the rate of change in the instrument score differed by treatment group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.7311, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000343, Standard Error of Mean 0.000996

3. Secondary Outcome: Defense and Veterans Pain Rating Scale
Description: 10-point scale to measure current pain intensity (past 24 hours) and pain interference (past 24 hours) with activity, sleep, mood, and stress.
  Higher Scores associated with more adverse pain-related patient reported outcomes.
  Pain Range: 0 - 10 Pain Interference with Activity Range: 0 - 10 Pain Interference with Sleep Range: 0 - 10 Pain Interference with Mood Range: 0 - 10 Pain Interference with Stress Range: 0 - 10
Time Frame: Baseline, month 1,2,4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Treatment Arm: Treatment Arm: MR is an user-driven, dyadic, self-care management program developed with National Institute of Mental Health (NIMH) funding (R43/44) for use by Veterans and their selected partners, individually or together, to reduce pain and distress and support physical, mental, and relationship health. MR was designed for Veterans who face obstacles accessing formal mental health services. It can also be used to complement formal services. MR is a patient-centered intervention, allowing users to determine the pace at which to proceed in each program component. MR Content. The program provides video and audio instruction in a set of 11 evidence-based wellness.
  Mission Reconnect: This four-year randomized controlled trial with one intervention arm and one wait-list control arm will utilize mixed methods to evaluate the effectiveness and perceived value of the MR program in relation to physical and psychological symptoms, global health, and social outcomes.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 141 | 136
units on a scale
  Overall Pain | 5.8062 [5.5361 to 6.0764] | 5.8431 [5.5821 to 6.1041]
  Pain Interference with Activity | 6.1319 [5.7757 to 6.4880] | 6.0125 [5.6658 to 6.3593]
  Pain Interference with Sleep | 5.9953 [5.5840 to 6.4066] | 5.7385 [5.3370 to 6.1400]
  Pain Interference with Mood | 6.1210 [5.7399 to 6.5021] | 5.9215 [5.5525 to 6.2905]
  Pain Interference with Stress | 6.0832 [5.6833 to 6.4831] | 5.8715 [5.4825 to 6.2605]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1622, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00241, Standard Error of Mean 0.001716
Statistical Analysis 2: Comparison: Treatment Arm vs Control Arm; Analysis performed on Pain Interference with Activity as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.2540, Mixed Models Analysis; Slope = -0.00235, Standard Error of Mean 0.002052
Statistical Analysis 3: Comparison: Treatment Arm vs Control Arm; Analysis performed on Pain Interference with Sleep as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0082, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00612, Standard Error of Mean 0.002297
Statistical Analysis 4: Comparison: Treatment Arm vs Control Arm; Analysis performed on Pain Interference with Mood as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0079, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00636, Standard Error of Mean 0.002378
Statistical Analysis 5: Comparison: Treatment Arm vs Control Arm; Analysis performed on Pain Interference with Stress as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1588, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00334, Standard Error of Mean 0.002367

4. Secondary Outcome: PTSD: Posttraumatic Checklist
Description: 20-item measure of PTSD symptoms Higher Scores associated with more adverse PTSD-related patient reported outcomes.
  Posttraumatic Stress Disorder Checklist (PCL-5) Range: 0 - 80
Time Frame: Baseline, month 1,2,4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 141 | 136
units on a scale | 43.5759 [40.8709 to 46.2810] | 41.5687 [38.9070 to 44.2304]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Analysis performed on PCL-5 Total Score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.4808, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00974, Standard Error of Mean 0.01379

5. Secondary Outcome: Quality of Life Short-form (SF12)
Description: 12-items to assess quality of life using physical status and mental health distress.
  Scores for the Mental Health and Physical Health domains range from 0 to 100, with higher scores indicating better physical and mental health functioning
Time Frame: Baseline, month 1,2,4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 141 | 136
units on a scale
  Physical Health Domain | 24.1845 [22.7008 to 25.6682] | 24.0067 [22.5597 to 25.4537]
  Mental Health Domain | 43.5871 [42.3829 to 44.7914] | 44.3803 [43.2200 to 45.5406]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Analysis performed on Physical Health Domain Score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.9692, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00033, Standard Error of Mean 0.008560
Statistical Analysis 2: Comparison: Treatment Arm vs Control Arm; Analysis performed on Mental Health Domain Score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0277, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.01738, Standard Error of Mean 0.007848

6. Secondary Outcome: Sleep Quality: Pittsburgh Sleep Quality Index (PSQI)
Description: 19 self-rated questions from which 7 component scores are calculated and summed into a global score to assess sleep quality in the past month.
  Each of the domain scores range from 0 (no difficulty) to 3 (severe difficulty).
  The global score ranges from 0 to 21. Higher scores indicate worse sleep quality.
Time Frame: Baseline, month 1,2,4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 141 | 136
units on a scale
  Pittsburgh Sleep Quality Index - Subjective sleep quality | 1.9406 [1.8262 to 2.0549] | 1.8286 [1.7189 to 1.9383]
  Pittsburgh Sleep Quality Index - Sleep latency | 2.0332 [1.8798 to 2.1867] | 2.0296 [1.8803 to 2.1790]
  Pittsburgh Sleep Quality Index - Sleep duration | 0.8399 [0.6662 to 1.0135] | 1.0488 [0.8852 to 1.2124]
  Pittsburgh Sleep Quality Index - Sleep efficiency | 0.3487 [0.2472 to 0.4502] | 0.3552 [0.2606 to 0.4498]
  Pittsburgh Sleep Quality Index - Sleep disturbance | 1.9855 [1.8898 to 2.0812] | 1.9507 [1.8589 to 2.0426]
  Pittsburgh Sleep Quality Index - Use of sleep medication | 1.9685 [1.7618 to 2.1751] | 1.9055 [1.7056 to 2.1054]
  Pittsburgh Sleep Quality Index - Daytime dysfunction | 1.7602 [1.6399 to 1.8806] | 1.6735 [1.5573 to 1.7897]
  Pittsburgh Sleep Quality Index - Global PSQI Score | 10.8145 [10.2417 to 11.3873] | 10.7561 [10.2006 to 11.3116]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Analysis performed on Total PSQI Score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.5642, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00188, Standard Error of Mean 0.003253
Statistical Analysis 2: Comparison: Treatment Arm vs Control Arm; Analysis performed on PSQI Subjective Sleep Quality Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.2438, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00092, Standard Error of Mean 0.000790
Statistical Analysis 3: Comparison: Treatment Arm vs Control Arm; Analysis performed on PSQI Sleep latency Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.7317, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000304, Standard Error of Mean 0.000885
Statistical Analysis 4: Comparison: Treatment Arm vs Control Arm; Analysis performed on PSQI Sleep duration Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.6393, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00062, Standard Error of Mean 0.001327
Statistical Analysis 5: Comparison: Treatment Arm vs Control Arm; Analysis performed on PSQI Sleep efficiency Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1995, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00112, Standard Error of Mean 0.000873
Statistical Analysis 6: Comparison: Treatment Arm vs Control Arm; Analysis performed on PSQI Sleep disturbance Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.2886, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00072, Standard Error of Mean 0.000675
Statistical Analysis 7: Comparison: Treatment Arm vs Control Arm; Analysis performed on PSQI Use of sleep medication Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1323, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.002048, Standard Error of Mean 0.001356
Statistical Analysis 8: Comparison: Treatment Arm vs Control Arm; Analysis performed on PSQI Daytime dysfunction Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.7923, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000209, Standard Error of Mean 0.000793

7. Secondary Outcome: Compassion for Self and Others Scales
Description: 26- item (CSS) and 21- item (COS) measures, that calculate an overall Compassion for Others score, an overall Compassion for Self score, and Compassion for Self subscale scores in the domains of Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, Overidentification.
  CSS subdomain scales and the total score (average of components) range from 0 - 5, with higher scores indicating higher self-compassion.
  COS score ranges from 0 - 7, with higher scores indicating higher compassion for others.
Time Frame: Baseline, month 1,2,4
Population: Multilinear model analyses were performed. Results provided are the Least Squares Mean and 95% C.I. for the two treatment arms. This is the least squares mean for the treatment variable averaged across all timepoints, after having controlled for other covariates. Instrument was administered only to Vets and Parts who had been activated in the protocol. Participants who opted out of responding to certain questions were not included in the analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm - Veteran | Treatment Arm - Partner | Control Arm - Veteran | Control Arm - Partner
Number analyzed (Participants) | 141 | 137 | 136 | 133
units on a scale
  Overall COS | 5.5055 [5.3181 to 5.6930] | 6.1296 [6.0026 to 6.2565] | 5.4667 [5.2829 to 5.6505] | 5.9148 [5.7919 to 6.0376]
  Overall CSS | 2.7177 [2.5843 to 2.8510] | 3.2624 [3.1368 to 3.3880] | 2.7983 [2.6662 to 2.9305] | 3.2908 [3.1662 to 3.4155]
  CSS, Self-kindness Subdomain | 2.5769 [2.4215 to 2.7323] | 3.2407 [3.0931 to 3.3882] | 2.7097 [2.5581 to 2.8613] | 3.2320 [3.0876 to 3.3765]
  CSS, Self-judgment Subdomain | 2.4873 [2.3297 to 2.6449] | 3.0189 [2.8580 to 3.1798] | 2.5104 [2.3560 to 2.6648] | 3.0766 [2.9186 to 3.2346]
  CSS, Common Humanity Subdomain | 2.7811 [2.6305 to 2.9317] | 3.2938 [3.1377 to 3.4498] | 2.9178 [2.7723 to 3.0634] | 3.4125 [3.2607 to 3.5642]
  CSS, Isolation Subdomain | 2.6541 [2.4834 to 2.8248] | 3.2216 [3.0588 to 3.3844] | 2.6762 [2.5089 to 2.8436] | 3.2205 [3.0610 to 3.3799]
  CSS, Mindfulness Subdomain | 3.0142 [2.8653 to 3.1630] | 3.5882 [3.4454 to 3.7310] | 3.1499 [3.0052 to 3.2946] | 3.5835 [3.4442 to 3.7228]
  CSS, Over-identification Subdomain | 2.7745 [2.6027 to 2.9463] | 3.2191 [3.0614 to 3.3768] | 2.8186 [2.6499 to 2.9874] | 3.2389 [3.0843 to 3.3936]
Statistical Analysis 1: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on COS Total Score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.6679, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00046, Standard Error of Mean 0.001074
Statistical Analysis 2: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 7, analysis 1]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1607, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.001083, Standard Error of Mean 0.000769
Statistical Analysis 3: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on CSS- Total as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1260, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000984, Standard Error of Mean 0.000640
Statistical Analysis 4: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on CSS Self-Kindness Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.3311, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000909, Standard Error of Mean 0.000933
Statistical Analysis 5: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on CSS Self-Judgment Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.2416, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.001041, Standard Error of Mean 0.000887
Statistical Analysis 6: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on CSS Common Humanity Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.3903, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00087, Standard Error of Mean 0.001016
Statistical Analysis 7: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on CSS Isolation Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.2131, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.001186, Standard Error of Mean 0.000950
Statistical Analysis 8: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on CSS Mindfulness Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1130, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.001485, Standard Error of Mean 0.000933
Statistical Analysis 9: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on CSS Over-identification Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0358, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.001983, Standard Error of Mean 0.000939
Statistical Analysis 10: Comparison: Treatment Arm - Partner vs Control Arm - Partner; Analysis performed on CSS- Total Score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.7027, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00019, Standard Error of Mean 0.000495
Statistical Analysis 11: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 7, analysis 4]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.2979, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000761, Standard Error of Mean 0.000730
Statistical Analysis 12: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 7, analysis 5]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.4278, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00063, Standard Error of Mean 0.000798
Statistical Analysis 13: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 7, analysis 6]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.9933, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.0000074, Standard Error of Mean 0.000877
Statistical Analysis 14: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 7, analysis 7]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1589, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00115, Standard Error of Mean 0.000816
Statistical Analysis 15: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 7, analysis 8]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.8875, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000109, Standard Error of Mean 0.000767
Statistical Analysis 16: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 7, analysis 9]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.6859, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00032, Standard Error of Mean 0.000780

8. Other Pre Specified Outcome: Depression: Beck Depression Inventory (BDI)
Description: 21-items, a widely used instrument for measuring depression. Respondents are asked to rate their symptoms and attitudes using a 4-point scale.
  Beck Depression Inventory (BDI) scores range from 0 to 63 with higher scores indicating more likely depression diagnosis, and higher prevalence of depression symptoms.
Time Frame: Baseline, month 1,2,4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 141 | 136
units on a scale | 26.2981 [24.0543 to 28.5420] | 24.6833 [22.4713 to 26.8952]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Analysis performed on BDI total score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1959, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.01408, Standard Error of Mean 0.01085

9. Other Pre Specified Outcome: Stress: Perceived Stress Scale (PSS)
Description: 10 Likert-scaled items, validated and widely used, to determine perceived stress levels.
  Perceived Stress Scale (PSS) scaled from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: Baseline, month 1,2,4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 141 | 136
units on a scale | 22.9251 [21.8127 to 24.0376] | 21.9134 [20.8220 to 23.0049]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Analysis performed on Perceived Stress Scale Score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1792, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00788, Standard Error of Mean 0.005845

10. Other Pre Specified Outcome: Revised Dyadic Adjustment Scale (RDAS)
Description: 14-item Likert-scaled instrument that contains domains for dyadic Consensus (sub-domain Decision Making, Values, and Affection), dyadic Satisfaction (sub-domain Stability and Conflict), and dyadic Cohesion (sub-domain Activities and Discussion).
  Scores on the Revised Dyadic Adjustment Scale (RDAS) range from 0 to 69 with higher scores indicating greater relationship satisfaction and lower scores indicating greater relationship distress.
Time Frame: Baseline, month 1,2,4
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm - Veteran | Control Arm - Veteran | Treatment Arm - Partner | Control Arm - Partner
Number analyzed (Participants) | 141 | 136 | 136 | 133
units on a scale
  Total RDAS | 46.5186 [44.7637 to 48.2734] | 47.8727 [46.1710 to 49.5745] | 48.4518 [46.9360 to 49.9676] | 48.4138 [46.9186 to 49.9091]
  Subdomain: Decision Making. Consensus Domain, RDAS | 7.4194 [7.1090 to 7.7298] | 7.5229 [7.2281 to 7.8177] | 7.6760 [7.4422 to 7.9098] | 7.7975 [7.5747 to 8.0202]
  Subdomain: Values. Consensus Domain, RDAS | 7.4926 [7.2021 to 7.7830] | 7.3515 [7.0774 to 7.6256] | 7.3577 [7.0990 to 7.6163] | 7.5449 [7.2967 to 7.7931]
  Subdomain: Affection. Consensus Domain, RDAS | 6.3686 [5.9426 to 6.7947] | 6.7036 [6.3005 to 7.1066] | 7.0612 [6.7448 to 7.3776] | 7.2958 [6.9897 to 7.6020]
  Total Consensus Domain, RDAS | 21.2171 [20.3318 to 22.1025] | 21.5715 [20.7299 to 22.4130] | 22.0963 [21.4122 to 22.7805] | 22.5988 [21.9356 to 23.2620]
  Subdomain: Stability. Satisfaction Domain, RDAS | 8.1158 [7.7955 to 8.4360] | 8.1900 [7.8844 to 8.4957] | 8.3706 [8.0901 to 8.6511] | 8.2289 [7.9520 to 8.5058]
  Subdomain: Conflict. Satisfaction Domain, RDAS | 6.5146 [6.2132 to 6.8161] | 6.5229 [6.2323 to 6.8136] | 6.4356 [6.1667 to 6.7045] | 6.3987 [6.1332 to 6.6643]
  Total Satisfaction Domain, RDAS | 14.6541 [14.1082 to 15.1999] | 14.7285 [14.2022 to 15.2547] | 14.8108 [14.3100 to 15.3117] | 14.6276 [14.1307 to 15.1244]
  Subdomain: Activities. Cohesion Domain, RDAS | 4.1842 [3.8649 to 4.5035] | 4.6511 [4.3443 to 4.9579] | 4.6317 [4.3504 to 4.9129] | 4.6058 [4.3346 to 4.8771]
  Subdomain: Discussion. Cohesion Domain, RDAS | 6.5337 [6.1557 to 6.9117] | 6.8995 [6.5375 to 7.2614] | 6.9106 [6.5682 to 7.2530] | 6.5975 [6.2667 to 6.9284]
  Total Cohesion Domain, RDAS | 10.7219 [10.0900 to 11.3537] | 11.5612 [10.9506 to 12.1718] | 11.5357 [10.9654 to 12.1060] | 11.2067 [10.6549 to 11.7586]
Statistical Analysis 1: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Total RDAS as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.8991, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.001320, Standard Error of Mean 0.01039
Statistical Analysis 2: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Decision Making Subdomain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.3711, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.002105, Standard Error of Mean 0.002349
Statistical Analysis 3: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Values Subdomain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.4280, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.001864, Standard Error of Mean 0.002348
Statistical Analysis 4: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Affection Subdomain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.9831, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00007, Standard Error of Mean 0.003205
Statistical Analysis 5: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Total Consensus Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.6320, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.003052, Standard Error of Mean 0.006364
Statistical Analysis 6: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Stability Subdomain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.9755, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000070, Standard Error of Mean 0.002259
Statistical Analysis 7: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Conflict Subdomain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.7584, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000560, Standard Error of Mean 0.001818
Statistical Analysis 8: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Total Satisfaction Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.9313, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000297, Standard Error of Mean 0.003444
Statistical Analysis 9: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Activities Subdomain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.5401, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00129, Standard Error of Mean 0.002097
Statistical Analysis 10: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Discussion Subdomain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.9421, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.000180, Standard Error of Mean 0.002471
Statistical Analysis 11: Comparison: Treatment Arm - Veteran vs Control Arm - Veteran; Analysis performed on Total Cohesion Domain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.7042, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00151, Standard Error of Mean 0.003983
Statistical Analysis 12: Comparison: Treatment Arm - Partner vs Control Arm - Partner; Analysis performed on Total RDAS Score as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0114, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.02128, Standard Error of Mean 0.008331
Statistical Analysis 13: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 2]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1358, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.002587, Standard Error of Mean 0.001727
Statistical Analysis 14: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 3]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.4354, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.001402, Standard Error of Mean 0.001796
Statistical Analysis 15: Comparison: Treatment Arm - Partner vs Control Arm - Partner; Analysis performed on AffectionSubdomain as outcome variable. Linear mixed models were constructed with fixed effects terms for the Tx group (MR vs. WC), time (continuous), and a Tx group x time interaction term to test whether the rate of change in the instrument score differed by Tx group. Random effects for the intercept and time were also included. The α p-value for statistical significance was set at 0.01. Borderline statistical significance was considered to be <0.1; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0070, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.005759, Standard Error of Mean 0.002113
Statistical Analysis 16: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 5]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0217, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.01037, Standard Error of Mean 0.004485
Statistical Analysis 17: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 6]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.7881, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = -0.00039, Standard Error of Mean 0.001461
Statistical Analysis 18: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 7]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0010, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.004717, Standard Error of Mean 0.001410
Statistical Analysis 19: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 8]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.0693, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.004393, Standard Error of Mean 0.002415
Statistical Analysis 20: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 9]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1184, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.002959, Standard Error of Mean 0.001887
Statistical Analysis 21: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 10]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1301, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.003436, Standard Error of Mean 0.002262
Statistical Analysis 22: Comparison: Treatment Arm - Partner vs Control Arm - Partner; [analysis description as in outcome 10, analysis 11]; Test type: Other — Treatment is compared against a Waitlist Control Group; p = 0.1049, Mixed Models Analysis — p value provided is for interaction term between Time (continuous) * Treatment group (MR vs. WC); Slope = 0.006022, Standard Error of Mean 0.003697

11. Other Pre Specified Outcome: MR Program Satisfaction Items
Description: 11 eleven-point Likert-type items (i.e., 0-10) assess satisfaction using MR components, whether they would recommend MR, and massage satisfaction. Higher scores refer to higher satisfaction with MR.
Time Frame: Month 4
Population: Instrument requests experiences with treatment. Instrument only administered to Veterans and Partners in the Treatment Arm who were activated in the protocol. Participants who opted out of responding to certain questions were not included in the analyses for the instrument.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment Arm - Veteran | Treatment Arm - Partner
Number analyzed (Participants) | 133 | 133
units on a scale
  Response to "I am satisfied with the Mission Reconnect program." | 8 [6 to 10] | 8 [7 to 10]
  Response to "I would recommend Mission Reconnect to other Veterans and their partners." | 9 [7 to 10] | 8 [7 to 10]
  Response to "I am satisfied with the "Connecting to Yourself" activities." | 8 [6.5 to 9.5] | 8 [7 to 10]
  Response to "I am satisfied with my ability to connect with myself." | 8 [6 to 9] | 8 [7 to 10]
  Response to "I am satisfied with the "Connecting with Quiet" activities." | 8 [6 to 10] | 8 [7 to 10]
  Response to "I am satisfied with my ability to connect with quiet." | 8 [6 to 10] | 8 [6 to 10]
  Response to "I am satisfied with the "Connecting with Your Partner" activities." | 8 [6 to 10] | 8 [6 to 10]
  Response to "I am satisfied with my ability to connect with my partner." | 8 [5 to 10] | 7.5 [6 to 10]
  Response to "I am satisfied with receiving massage from my partner." | 8 [6 to 10] | 9 [6 to 10]
  Response to "I am satisfied with my ability to give my partner massage." | 8 [5 to 10] | 8 [7 to 10]
  Response to "I am satisfied with the Mission Reconnect Support Materials activities." | 8 [6 to 10] | 8 [6 to 10]

12. Other Pre Specified Outcome: MR Program Utilization
Description: Treatment group: weekly report 11-items will assess frequency of use and compliance of the MR mind/body & massage practices. Measure calculated in number of minutes per week the participant performed the activity.
Time Frame: Month 4
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: minutes per week
Arm/Group | Treatment Arm - Veteran | Treatment Arm - Partner
Number analyzed (Participants) | 133 | 133
minutes per week
  Utilization in the "Connecting with Yourself" Domain | 30 [0 to 110] | 55 [15 to 98]
  Utilization in the "Connecting with the Quiet" Domain | 40 [0 to 98] | 42 [10 to 95]
  Utilization in the "Connecting with your Partner" Domain | 60 [0 to 240] | 43 [9 to 140]
  Total Utilization | 201 [0 to 565] | 190 [70 to 360]

ADVERSE EVENTS:
Time Frame: Baseline (before the start of the study activities) and 1, 2 & 4 months after study activities)
Description: While all participants are given a baseline coverage of resources to deal with suicidal ideation, domestic violence issues, and/or severe depression/mental health issues, the Veteran participants are also directly asked at Baseline and at the monthly time points if they specifically have suicidal ideation. An affirmative response of any suicidal ideation with intent and/or plan of action.
Arm/Group | Treatment Arm - Veteran | Treatment Arm - Partner | Control Arm - Veteran | Control Arm - Partner
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/198 | 0/168 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/198 | 0/168 | 0/168
Other Adverse Events (participants affected / at risk) | 7/196 | 0/198 | 7/168 | 0/168
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm - Veteran (N=196) | Treatment Arm - Partner (N=198) | Control Arm - Veteran (N=168) | Control Arm - Partner (N=168)
Suicide Ideation (Social circumstances) | 7 (16) | 0 (0) | 7 (8) | 0 (0) — Participants reported suicide ideation as part of Patient Reported Outcomes. All Suicide Ideation was escalated to the Veteran's Mental Health provider as per protocol and VA policies.

LIMITATIONS AND CAVEATS:
Demographics were calculated from study dyads who were successfully activated in the study. Successful activation required both Veteran and Partner of a dyad to complete all Baseline measures. Certain dyads consisted of individuals where one partner completed Baseline data collection before either withdrawing or being Lost to Follow Up (unrelated to study activities). Their data, as per study protocol, were still included in the data models, but were not included in Demographic summaries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT03593772/Prot_SAP_ICF_000.pdf